CLINICAL TRIAL: NCT01242566
Title: Phase II Trial of Temozolomide in Elderly Patients With Glioblastoma and Poor Performance Status (KPS<70).
Brief Title: Temozolomide in Elderly Patients With KPS < 70
Acronym: TAG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association de Neuro-Oncologues d'Expression Francaise (Other)
Responsible Party: Isabelle Brindel, Department Clinical Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P060102
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Primary Brain Tumor; Glioblastoma
Keywords: Temozolomide; Elderly; Glioblastoma; Karnofsky performance score (KPS)
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- temozolomide (Experimental): Administration of temozolomide 150-200 mg/m2/day for 5 consecutive days every 4 weeks for a maximum of 12 cycles or until disease progression or prohibited toxicity
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — orally 150-200 mg/m2/day for 5 consecutive days every 4 week
  Other Names: Temodar, Temodal

SUMMARY:
The management of glioblastoma in elderly patients with poor performance status (KPS<70) is unsettled. This single arm phase 2 trial trial was designed to evaluate the efficacy and safety of temozolomide alone in this population

DETAILED DESCRIPTION:
This trial was conducted to evaluate the efficacy, in terms of survival and quality of life, and safety of up-front temozolomide in elderly GBM patients with poor performance status.

Patients of 70 years of age or older were eligible to participate in this prospective non-randomised multicentric phase II study if they had newly diagnosed and histologically proven glioblastoma on the basis of the WHO classification, and a postoperative KPS between 30 and 60.

Treatment consisted of temozolomide 150-200 mg/m2/day for 5 consecutive days every 4 weeks for a maximum of 12 cycles or until disease progression or prohibited toxicity.

Patients were assessed at least every month by means of physical and neurological examinations, KPS, health-related EORTC questionnaires (QLQ-C30 and QLQ-BN20), and MMSE. Complete blood counts and blood chemistry were drawn before each temozolomide cycle; the earlier were also checked every 10 days during the first 2 cycles and every 2 weeks afterwards. CT or MRI studies were repeated every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed supratentorial glioblastoma
* Baseline contrast-enhanced CT or gadolinium-enhanced MRI study performed within the first 4 days from resection or within the first 4 weeks from diagnostic biopsy
* Patients aged 70 years or older
* KPS above 30 and below 70
* Life expectancy higher than 4 weeks
* Clinical examination at baseline
* Affiliation to Social Security or mandatory beneficiary
* Patient being informed and obtention of written informed consent

Exclusion Criteria:

* Prior surgical resection dated more than 1 month before inclusion
* Prior brain radiotherapy or chemotherapy
* Severe underlying disease which could interfere with survival
* History of hypersensibility reaction on temozolomide components
* Severe bone marrow hypoplasia
* Aspartate aminotransferase or alanine aminotransferase more than 3 times the upper limit of normal
* Absolute neutrophil count < 1.5x109 cells per liter
* Platelet count < 100x109 cells per liter
* Hemoglobin < 9 g/dl
* Neuroimaging baseline examination performed beyond the first 4 days from resection or beyond the first 4 weeks from diagnostic biopsy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2007-07; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | 12 months

SECONDARY OUTCOMES:
Progression-free survival | 12 months
adverse events | 12 months
  term, grade, frequency
Health-related quality of life | 12 months
  KPS and EORTC questionnaires (QLQ-C30 and QLQ-BN20)
Cognitive functioning | 12 months
  characterized by MMSE
Efficacy according to MGMT Promoter methylation status | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: DELATTRE Jean-Yves, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pitie salpetriere hospital, Paris, France